CLINICAL TRIAL: NCT06808347
Title: Difference in Serum Estrogen Level Based on Methods of Vaginal Estrogen Application (fingertip Vs Applicator Use) in Post-menopausal Women
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRNMMC-2023-0432
Record Dates: First submitted 2024-12-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Postmenopausal Atrophic Vaginitis; Genitourinary Syndrome of Menopause
MeSH Terms: conditions — Atrophic Vaginitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vaginal estrogen application in post-menopausal women by fingertip use (Active Comparator): will include post-menopausal women who are applying the vaginal estrogen cream by using their fingertip
  Interventions: Drug: application of the vaginal estrogen cream
- vaginal estrogen application in post-menopausal women by applicator use (Active Comparator): will include post-menopausal women who are applying the vaginal estrogen cream by using the applicator
  Interventions: Drug: application of the vaginal estrogen cream

INTERVENTIONS:
Drug: application of the vaginal estrogen cream — patients will apply the vaginal estrogen cream

SUMMARY:
Study the change in serum estrogen level based on the method of vaginal cream application (applicator vs fingertip application) and Measure patient satisfaction with vaginal estrogen cream application based on the method of application using a validated patient questionnaire (Likert scale).

DETAILED DESCRIPTION:
Describe step-by-step how the study will be conducted from beginning to end All women who are over the age of 18 who meet criteria for post-menopausal state, with symptoms of genitourinary syndrome of menopause, who qualify for local vaginal estrogen therapy and who are receiving care at Walter Reed National Military Medical Center (WRNMMC) in the Gynecological Surgery and Obstetrics department clinic will be eligible for the study.

All study participants will undergo a complete intake assessment to include a history, medication reconciliation, allergies verification, physical exam, and counseling on treatment modalities for genitourinary syndrome of menopause to include lubrication, vaginal moisturizers, non-hormonal treatments, vaginal estrogen treatment and laser therapy. The AUGS handout about vaginal estrogen therapy will be given to patients. Patients desiring treatment with vaginal estrogen therapy and meeting our inclusion and exclusion criteria will be offered enrollment in this study.

Enrollment will be done by the research team consisting of the clinician. No patient will be pressured or coerced into participating in the study. During the enrollment visit, participants will be consented for participation in the study and asked to complete a demographics data sheet and a female sexual function index questionnaire.

The statistician will make randomized assignments which will be concealed in sequentially numbered opaque envelopes which will be opened on the day of enrollment by the treatment provider. The envelop will reveal the method of application of the vaginal estrogen cream (applicator vs fingertip application). The provider will then reveal the allocation treatment group to the patient. The vaginal estradiol cream Estrace (chosen due to lower cost than other vaginal estrogen formulations) will then be provided to the patient. If the patient is allocated to the applicator group, a demonstration of the application will be completed in clinic using a vaginal model and a sample applicator. If the patient is allocated to the fingertip application, a demonstration of the application will be completed in clinic using a vaginal model. Printed information about each method of application will be provided to patients in both groups. Serum estrogen level will be drawn in the lab during this visit as a baseline measure for future comparison (the patient will be sent to the lab for the serum estrogen level to be drawn).

Standard of care treatment: 0.5g of the vaginal estrogen cream is inserted using the applicator into the vagina once a day for 2 weeks, followed by 3 times per week.

The research component will be to insert a pea size amount of the estrogen cream into the vagina using the index finger (finger application) once a day for 2 weeks, followed by 3 times per week.

The patient satisfaction questionnaires, blood draws to check the serum estrogen levels, and the 6-10 week follow up visit are not standard of care and will be part of our research component done for the purpose of this study. our research aims to study the difference in serum estrogen level based on the method of application of the vaginal estrogen cream: using the applicator ( which is standard of care) vs using fingertip application of the cream into the vagina (research component).

Patients will be instructed to apply the vaginal estrogen cream daily for 2 weeks, followed by 3 times per week for an additional 4-8 weeks (total 6-10 weeks). Patients will be offered an in person follow up appointment at 6-10 weeks after starting the vaginal estrogen cream. they can also be offered a virtual visit via telephone or electronic health record patient portal. if they elect to have a virtual visit, they will be asked to drop off their vaginal estrogen tube in a drop box in clinic for the tube to be weighed for compliance and will also be asked to go to the lab to have their blood drawn to check the serum estrogen level.

During the in-person follow up visit, the vaginal estradiol cream will be measured by weighing the tube to confirm patient's compliance with the treatment. The patient will be asked to complete a second female sexual function index questionnaire to compare to the baseline questionnaire, as well as a Likert scale questionnaire to evaluate satisfaction with the application method. Serum estrogen levels will be drawn again by having the patient go to the lab to compare to baseline as well (to the initial serum level that was drawn during the initial visit).

After study completion, patients are given the option to continue using the vaginal estrogen cream indefinitely or to discontinue it if they are not satisfied with the treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients who are postmenopausal for at least 1 year (since their last menses)
* patients who qualify for treatment with vaginal estrogen cream and are willing to complete the treatment
* English speaking patients
* patients should be able to self-apply the vaginal estrogen cream using the applicator method and the fingertip application
* Patients who are surgically menopausal
* Military healthcare beneficiary status

Exclusion Criteria:

* pre and perimenopausal women
* contraindication to estrogen therapy (Deep vein thrombosis, history or active cancer)
* women who are not able to self apply the vaginal estrogen cream
* vaginal bleeding of unknown origin
* women currently on hormone replacement therapy or vaginal estrogen therapy

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Measure the change in the level of serum estrogen in postmenopausal women based on the method of application of the estrogen cream (fingertip vs applicator use). | 6-8 weeks

SECONDARY OUTCOMES:
Measure patient satisfaction with vaginal estrogen cream application based on the method of application using a validated patient questionnaire (Likert scale). | 6-8 weeks
Measure improvement in sexual dysfunction with application of the vaginal estrogen cream based on the method of application using a validated patient questionnaire (Female sexual function index). | 6-8 weeks

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code